CLINICAL TRIAL: NCT04374981
Title: Effect of Pineapple Juice on the Pharmacokinetics of Celecoxib and Montelukast in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Sally Helmy, PhD, CPHQ, Associate professor, Damanhour University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CMP
Record Dates: First submitted 2020-04-24; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Food-drug Interaction
MeSH Terms: interventions — Celecoxib; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celecoxib (Experimental): Twelve healthy male subjects participated in this arm under fasting condition. A randomized, open-label, 2-way crossover study design with 2-week washout period between treatments was used. Participants received a single oral dose of celecoxib tablets (100mg) after pre-treatment with 250ml of either pineapple juice or water (control) for four consecutive days before the beginning of the study.
  Interventions: Drug: Celecoxib 100mg
- Montelukast (Experimental): Twelve healthy male subjects participated in this arm under fasting condition. A randomized, open-label, 2-way crossover study design with 2-week washout period between treatments was used. Participants received a single oral dose of Montelukast tablets (10mg) after pre-treatment with 250ml of either pineapple juice or water (control) for four consecutive days before the beginning of the study.
  Interventions: Drug: Montelukast 10mg

INTERVENTIONS:
Drug: Celecoxib 100mg — Tablets
  Arms: Celecoxib
Drug: Montelukast 10mg — Tablets
  Arms: Montelukast

SUMMARY:
Pineapple (Ananas comosus) is a tropical fruit that is rich in antioxidents, enzymes and vitamins. It is used worldwide due to their anti-inflammatory and analgesic properties. The effect of pineapple Juice on the Pharmacokinetics of celecoxib and montelukast in Humans was studied.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (body mass index between 21 to 25 kg/m2).

Exclusion Criteria:

* Smokers.
* Drug abuse.
* Abnormal level of kidney or liver functions.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | 12 weeks
Time to reach plasma peak concentration [Tmax] | 12 weeks
Time to reach maximum plasma concentration [Tmax] | 12 weeks
The area under the concentration-time curve from zero to infinity (AUC0-∞) | 12 weeks
The terminal elimination half-life (t1/2) | 12 weeks

SECONDARY OUTCOMES:
Clearance (CLT/F) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sally Helmy, PhD, Principal Investigator — Damanhour University
Locations (1):
- Faculty of Pharmacy-Damanhour University., Damanhūr, Egypt

IPD SHARING:
Plan to Share IPD: Yes